CLINICAL TRIAL: NCT05433467
Title: The Feasibility of CT-guided Localization for Micro Hepatocellular Carcinoma Before Surgical Resection
Brief Title: CT-guided Localization for Micro Hepatocellular Carcinoma Before Surgical Resection
Acronym: CTMH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Northern Jiangsu People's Hospital (Other)
Responsible Party: Principal Investigator, Guo-Qing Jiang, Clinical Professor, Northern Jiangsu People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YZUC-012
Record Dates: First submitted 2022-06-21; First posted 2022-06-27 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Cirrhosis, Liver; Hepatocellular Carcinoma
Keywords: Cirrhosis; hepatocellular carcinoma; localization needle
MeSH Terms: conditions — Liver Cirrhosis; Carcinoma, Hepatocellular; Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CT-guided localization for micro hepatocellular carcinoma before surgical resection (Experimental): fter preoperative preparation was completed, on the day of surgery, disposable pulmonary nodular localization needle (Ningbo Sonjiecang Biological Technology Co., LTD., Model: SS510-10) was used for the localization of micro hepatocellular carcinoma that could be found by preoperative CT enhancement or MRI. After the micro hepatocellular carcinoma was located under the guidance of CT, and then the patient was sent to the operating room. During the operation, the lesion was removed according to the tail line of the positioning needle and the position of the positioning needle.
  Interventions: Procedure: CT-guided localization for micro hepatocellular carcinoma before surgical resection

INTERVENTIONS:
Procedure: CT-guided localization for micro hepatocellular carcinoma before surgical resection — After preoperative preparation was completed, on the day of surgery, disposable pulmonary nodular localization needle (Ningbo Sonjiecang Biological Technology Co., LTD., Model: SS510-10) was used for the localization of micro hepatocellular carcinoma that could be found by preoperative CT enhancement or MRI. After the micro hepatocellular carcinoma was located under the guidance of CT, and then the patient was sent to the operating room. During the operation, the lesion was removed according to the tail line of the positioning needle and the position of the positioning needle.

SUMMARY:
In this project, the preoperative anatomical location of micro hepatocellular carcinoma under the guidance of CT can provide guidance for accurate surgical resection. It may also shorten the operation time and reduce intraoperative bleeding.

DETAILED DESCRIPTION:
General and basic information of the patients included in the study was collected. After preoperative preparation was completed, on the day of surgery, disposable pulmonary nodular localization needle (Ningbo Sonjiecang Biological Technology Co., LTD., Model: SS510-10) was used for the localization of micro hepatocellular carcinoma that could be found by preoperative CT enhancement or MRI. After the micro hepatocellular carcinoma was located under the guidance of CT, and then the patient was sent to the operating room. During the operation, the lesion was removed according to the tail line of the positioning needle and the position of the positioning needle.

ELIGIBILITY:
Inclusion Criteria:

1. Be at least 18 years old and give informed consent to participate in the study
2. A preoperative (clinical, radiological, or histological) diagnosis of cirrhosis of the liver due to any cause.
3. micro hepatocellular carcinoma (diameter less than 1cm).
4. Preoperative CT plain scan could not find the lesion, and preoperative B-ultrasound could not find the lesion.
5. Preoperative CT enhancement or MRI can detect the lesion.

Exclusion Criteria:

1. Child-Pugh grade C
2. Uncontrolled Hypertension
3. Severe lung dysfunction
4. Severe cardiac dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
The position of the needle | During operation
  The distance (mm) of the needle to the edge of hepatocellular carcinoma

SECONDARY OUTCOMES:
Operation time | During operation
  The length of operation time (min)
Intraoperative bleeding | During operation
  The volume of intraoperative bleeding (ml)

CONTACTS AND LOCATIONS:
Overall Officials: Guo-Qing Jiang, MD, Study Chair — Clinical Medical College, Yangzhou University
Locations (1):
- Clinical Medical College, Yangzhou University, Yangzhou, Jiangsu, China